CLINICAL TRIAL: NCT01867996
Title: To Evaluate the Pharmacokinetics, Safety and Tolerability of Retosiban (GSK221149) Co-administered With EFAVIRENZ
Brief Title: A Study to Evaluate the Pharmacokinetics, Safety and Tolerability of Retosiban (GSK221149) When Dosed With Efavirenz (EFZ)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 116073
Record Dates: First submitted 2013-05-30; First posted 2013-06-04 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Obstetric Labour, Premature
Keywords: Retosiban, Efavirenz, Induction
MeSH Terms: conditions — Premature Birth | interventions — GSK221149A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Retosiban and EFZ (Experimental): All subjects will receive on Day 1, a 6 mg bolus of retosiban for 5 min, followed by a 6 mg/hr infusion for 12 hrs. On Day 2 a washout day will occur. On Days 3-17, subjects will receive EFZ 600 mg OD dose of in the evening. On Day 18, subjects will receive a 6 mg bolus of retosiban for 5 mins, followed by a 6 mg/hr infusion for 12 hrs plus a 600 mg dose of EFZ.
  Interventions: Drug: Retosiban; Drug: EFZ 600 mg

INTERVENTIONS:
Drug: Retosiban — Retosiban will be supplied as clear colorless solution for infusion (300 mg in 20 mL via). Subject will receive loading dose of 6 mg over 5 min infusion followed by 6 mg/hour infusion for 12 hrs on Day 1 and Day 18.
Drug: EFZ 600 mg — EZF 600 mg will be supplied as a yellow, capsular-shaped, film-coated tablet. Subjects will receive EFZ 600mg OD in the evening from Day 3 till Day 18.

SUMMARY:
This will be a randomized single sequence open label study. This study is designed to determine if chronic dosing with efavirenz (EFZ) will have an effect on the pharmacokinetics (PK) of intravenously-administered retosiban in healthy volunteers. The study consists of screening (28 days), treatment (1 dosing session) and follow-up (7 to 14 days) period, and the total duration of study participation for each subject will be approximately 8 weeks. During the treatment period, subjects will be admitted to the clinical research unit the day before dosing (Day 1) and will remain until completion of the last assessment on Day 20. All subjects will receive on Day 1, a 6 milligrams (mg) bolus of retosiban for 5 minutes (min), followed by a 6 mg/hour (hr) infusion for 12 hrs. On Day 2, a washout day will occur. On Days 3-17, subjects will receive EFZ 600 mg once daily in the evening. On Day 18, subjects will receive a 6 mg bolus of retosiban for 5 mins, followed by a 6 mg/hr infusion for 12 hrs plus a 600 mg dose of EFZ.

ELIGIBILITY:
Inclusion Criteria:

* Male/females aged between 18 and 45 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the Investigator in consultation with the GlaxoSmithKline (GSK) Medical Monitor agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >=50 kilogram (kg) and body mass index within the range 19-29.9 kg/m^2.
* A female subject is eligible to participate if she is of: Child-bearing potential with negative pregnancy test as determined by serum human chorionic gonadotrophin (hCG) test at screening or prior to dosing; AND Agrees to use the contraception methods for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until the follow-up visit; OR has only same-sex partners, when this is her preferred and usual lifestyle.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form
* Alanine aminotransferase (ALT), alkaline phosphatase and bilirubin <=1.5 x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Based on averaged corrected QT interval (QTc) values of triplicate electrocardiograms obtained over a brief recording period: QTc < 450 milliseconds (msec); or QTc < 480 msec in subjects with Bundle Branch Block.

Exclusion Criteria:

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of regular alcohol consumption within 6 months of the study defined as: For United States (US) sites: an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 gram of alcohol: 12 ounces (360 milliliter [mL]) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Has active suicidal plan/intent or has had active suicidal thoughts in the past 6 months. Has history of suicide attempt in the last 2 years or more than 1 lifetime suicide attempt.
* Subjects with a history of seizures will be excluded from this trial.
* Subjects with a history of severe or serious psychiatric disease requiring hospitalization, history of social ideation or attempt, or on ongoing psychiatric treatment will be excluded from this study.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* A positive pre-study drug/alcohol screen.
* A positive test for Human Immunodeficiency Virus (HIV) antibody.
* Pregnant females as determined by positive serum hCG test at screening or prior to dosing.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Lactating females.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2013-06-11 (Actual); Primary Completion 2013-09-26 (Actual); Study Completion 2013-09-26 (Actual)

PRIMARY OUTCOMES:
Plasma GSK221149 (parent) and GSK2847065 (metabolite) PK parameters of AUC, Cmax and CL. | 0, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 10, 12, 14, 16, 18, and 24 hours (hrs) after the start of the infusion on Day 1 and Day 18.
  The following PK parameters will be determined after administration of GSK221149 with and without EFZ 600 mg: Area under the plasma concentration-time curve (AUC)- from time zero to time t [AUC(0-t)] and from time zero extrapolated to infinite time [AUC(0-infinity)], maximum observed plasma concentration (Cmax) and clearance (CL). CL will be calculated for parent only.

SECONDARY OUTCOMES:
Safety and tolerability of administration of GSK221149 with and without EFZ 600 mg as assessed by adverse event, concurrent medication review, clinical laboratory tests, ECG, and vital signs measurements. | Up to 8 Weeks
  Clinical laboratory tests will include hematology, clinical chemistry and urinalysis parameters. Triplicate 12-lead ECGs will be obtained at the screening visit. Single 12-lead ECGs will be obtained at other time points during the study. Vital sign measurements will include systolic and diastolic blood pressure and pulse rate.
Plasma GSK221149 and GSK2847065 PK parameters of tmax, tlag and t1/2. | 0, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 10, 12, 14, 16, 18, and 24 hours (hrs) after the start of the infusion on Day 1 and Day 18.
  The following PK parameters will be determined after administration of GSK221149 with and without EFZ 600 mg: time to Cmax (tmax), lag time (tlag), and terminal phase half-life (t1/2). The terminal half-life (t1/2) is defined as the time required for the plasma concentration of drug to reach half of its original concentration.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 116073 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/116073?search=study&study_ids=116073#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 116073 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116073 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116073 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116073 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116073 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116073 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116073 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register